CLINICAL TRIAL: NCT00002831
Title: A Phase I/II Study of High-Dose Deoxyazacytidine, Busulfan, and Cyclophosphamide With Allogeneic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Chronic Myelogenous or Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM94-064; P30CA016672 (NIH); MDA-DM-94064 (Other: UT MD Anderson Cancer Center); NCI-G96-0999; CDR0000065033 (Registry Identifier: NCI's PDQ Database)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; Decitabine; Methotrexate; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deoxyazacytidine + Busulfan + Cyclophosphamide (Experimental): Deoxyazacytidine + Busulfan + Cyclophosphamide With Allogeneic Stem Cell Transplantation
  Interventions: Biological: Filgrastim; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Decitabine (DAC); Drug: Methotrexate; Drug: Methylprednisolone; Drug: Tacrolimus; Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Filgrastim — Subcutaneously (SQ) daily every 12 hours starting 2-4 days prior to the first stem cell collection and before DAC infusion.
  Other Names: C-CSF; Neupogen
Drug: Busulfan — Administered orally every 6 hours on consecutive days -6 through -4.
  Other Names: Busulfex; Myleran
Drug: Cyclophosphamide — Given intravenously (IV) over 1 hour on consecutive days -3 and -2.
  Other Names: Cytoxan; Neosar
Drug: Cyclosporine — Patients intolerant to tacrolimus receive cyclosporine IV beginning on day -2, then orally following tolerance and engraftment.
  Other Names: Sandimmune; CYA; Cyclosporin A
Drug: Decitabine (DAC) — IV over 4 hours on days -8 and -7.
  Other Names: Dacogen
Drug: Methotrexate — Given intrathecally or intraventricularly monthly, beginning on the second month through the eighth month of treatment.
Drug: Methylprednisolone — Given according to clinical grade of GVHD procedures.
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
Drug: Tacrolimus — IV beginning one day before stem cell infusion, then orally following tolerance to tacrolimus.
  Other Names: Prograf
Procedure: Allogeneic Bone Marrow Transplantation — Infusion of stem cells on Day 0.
  Other Names: ABMT
Procedure: Peripheral Blood Stem Cell Transplantation — Stem cell infusion on Day 0.
  Other Names: PBSCT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of high-dose chemotherapy plus peripheral stem cell transplantation in treating patients with chronic myelogenous or acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of decitabine in combination with busulfan and cyclophosphamide in patients with hematologic malignancies. II. Establish the pharmacokinetics of decitabine and busulfan in this patient population. III. Determine the effectiveness of this combination in achieving durable complete remission in patients with chronic myelogenous leukemia (CML) in blast crisis or acute myelogenous leukemia (AML) in relapse undergoing allogeneic stem cell transplantation.

OUTLINE: In cohorts of 3, patients receive escalating doses of decitabine (DAC) IV over 4 hours on days -8 and -7. Busulfan is administered orally every 6 hours on consecutive days -6 through -4. Cyclophosphamide is given by vein (IV) over 1 hour on consecutive days -3 and -2. The maximum tolerated dose of DAC is defined as the dose at which 2 patients experience dose limiting toxicity. Donors receive filgrastim subcutaneously (SQ) daily every 12 hours starting 2-4 days prior to the first stem cell collection and before DAC infusion. Leukapheresis is conducted daily. If insufficient number of cells are collected, blood marrow is harvested for supplementation. Stem cells are infused on day 0. For graft vs host disease prophylaxis (GVHD), patients receive tacrolimus IV beginning one day before stem cell infusion, then orally following tolerance to tacrolimus. Patients intolerant to tacrolimus receive cyclosporine IV beginning on day -2, then orally following tolerance and engraftment. All patients receive methylprednisolone given according to clinical grade of GVHD procedures. For CNS prophylaxis, methotrexate is given intrathecally or intraventricularly monthly, beginning on the second month through the eighth month of treatment. Allogeneic patients are followed until the end of 1 year.

PROJECTED ACCRUAL: An estimated 30 allogeneic recipients will be recruited in 2 years for the expected study duration of 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute leukemia past first remission or induction failure Chronic myelogenous leukemia in accelerated phase or blast crisis

PATIENT CHARACTERISTICS: Age: 15 to 55 Performance status: Zubrod 0-2 Life expectancy: Life expectancy not severely limited by concurrent illness Hematopoietic: Not specified Hepatic: No evidence of chronic active hepatitis or cirrhosis Bilirubin no greater than 2 times upper limit of normal SGPT no greater than 4 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: Left ventricular ejection fraction at least 50% No uncontrolled arrhythmias or symptomatic cardiac disease Pulmonary: FEV1, FVC, and DLCO at least 50% No symptomatic pulmonary disease Other: Related donor who is HLA-identical required No effusion or ascites greater than 1 L prior to drainage HIV negative Not pregnant No active CNS disease

PRIOR CONCURRENT THERAPY: Not specified

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 1995-08-01 (Actual); Primary Completion 2002-12-31 (Actual); Study Completion 2002-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Study Duration 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States